CLINICAL TRIAL: NCT01421004
Title: A Phase I, Open-label, Multi-center, Randomized, Crossover Study to Assess the Bioequivalence of 2 Formulations of TKI258, FMI Capsule and FMI Tablet, in Patients With Advanced Solid Tumors
Brief Title: Bioequivalence of 2 Formulations of TKI258 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258A2128
Record Dates: First submitted 2011-08-11; First posted 2011-08-22 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2015-01

CONDITIONS: Advanced Solid Tumors; Excluding Breast Cancer
Keywords: cancer; tumors; phase I; crossover; bioequivalence
MeSH Terms: conditions — Neoplasms | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

ARMS (2):
- 500 mg FMI capsule + 250 mg FMI tablet (Experimental): BE phase sequence 1= 3 weeks on FMI capsule then 1 week on FMI tablet
  Interventions: Drug: TKI258
- 500 mg TKI258 FMI capsule +250 mg FMI tablet (Experimental): BE phase sequence 2= 3 weeks on FMI tablet then 1 week on FMI capsule
  Interventions: Drug: TKI258

INTERVENTIONS:
Drug: TKI258
  Other Names: dovitinib

SUMMARY:
This is a multi-center, open-label, two way crossover study designed to test the bioequivalence of 2 different oral forms of TKI258, FMI capsule and FMI tablet in patients with advanced solid tumors, excluding breast cancer. The aim of this test is to demonstrate that those 2 formulations are considered to be the same for all intents and purposes by making sure they are acting on the body with the same strength and are absorbed in similar amounts by the body. During the bioequivalence phase, patients will take orally at a daily dose of 500 mg one formulation of TKI258 during the first 3 weeks of treatment on a 5 days on/2days off dosing schedule, after which time, patients will switch to the alternate formulation for one additional week. After the bioequivalence phase, all patients may continue to take orally at a daily dose of 500 mg only TKI258 FMI capsule formulation until disease progression (assessed by RECIST 1.1), unacceptable toxicity, death or discontinuation from the study treatment for any other reason.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a histopathologically or cytopathologically confirmed diagnosis of an advanced solid tumor, excluding breast cancer, who have progressed despite standard therapy, or for which no standard therapy exists
2. ECOG performance status (PS) 0, 1 or 2
3. Patients must meet protocol-specified laboratory values

Exclusion Criteria:

1. Patients with brain metastases
2. Patients who have concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study
3. Patients who have not recovered from previous anti-cancer therapies
4. Patients who are expected to receive any prohibited medications during the bioequivalence phase of the study
5. Female patients who are pregnant, breast feeding
6. Fertile male or women of child-bearing potential not willing to use two highly effective methods of contraception

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2011-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Composite of Pharmacokinetics of TKI258, FMI capsule (supplied in 100 mg strength) and FMI tablet (supplied in 250 mg strength), in patients with advanced solid tumors, excluding breast cancer based on PK parameters AUClast and Cmax | 9 days

SECONDARY OUTCOMES:
Frequency of Adverse Events in patients treated with TKI258 on a 5 days on/2 days off dosing schedule in patients with advanced solid tumors, excluding breast cancer | up to 30 days after the last dose of study drug
Preliminary evidence of anti-tumor activity based on RECIST criteria of TKI258 in patients with advanced solid tumors, excluding breast cancer | Every 8 weeks until progression of disease

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartitis Pharmaceuticals, Study Director — Novartitis Pharmaceuticals
Locations (14):
- United States (14):
  - City of Hope National Medical Center SC-2, Duarte, California
  - University of California at Los Angeles UCLA LeConte Location, Los Angeles, California
  - University of California San Francisco UCSF (SC), San Francisco, California
  - Florida Cancer Specialists Sarasota Office, Fort Myers, Florida
  - Rush University Medical Center Rush 3, Chicago, Illinois
  - Washington University School of Medicine SC, St Louis, Missouri
  - Montefiore Medical Center Montefiore Medical Center (SC), The Bronx, New York
  - University of Oklahoma Health Sciences Center OUHSC - SC, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute Sarah Cannon Research (SC), Nashville, Tennessee
  - Sammons Cancer Center - Texas Oncology SC-2, Dallas, Texas
  - Cancer Therapy & Research Center / UT Health Science Center InstituteForDrugDevelopment(5), San Antonio, Texas
  - University of Utah / Huntsman Cancer Institute Huntsman, Salt Lake City, Utah
  - University of Wisconsin Univ Wisc, Madison, Wisconsin

REFERENCES:
- See also: Results for CTKI258A2128 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13570